CLINICAL TRIAL: NCT05852210
Title: The Correlation of Thermal FLIR Imaging and Severity Score in Patients With Newly Diagnosed CRPS
Brief Title: Forward Looking InfraRed Imaging and Severity Score in Complex Regional Pain Syndrome
Acronym: FLIR
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2175
Record Dates: First submitted 2023-03-09; First posted 2023-05-10 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-01

CONDITIONS: CRPS (Complex Regional Pain Syndromes)
Keywords: Infrared; CRPS
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infrared CRPS Group: This group includes people who have recently been diagnosed with CRPS type 1. Participants in the Infrared group will have their feet photographed using a:
  * FLIR T420 or T62101 camera with 320*240 resolution.
  * Each image will be captured at a perpendicular angle with a 1-inch gap on all four sides.
  * The patients' feet will be separated from the background using a Myler blanket.
  * The camera will be normalized to the temperate range of 15°C minimum and 40°C maximum.
  * Patients will complete questionnaires about the severity of their CRPS and their pain levels.
  Interventions: Other: Infrared Imaging

INTERVENTIONS:
Other: Infrared Imaging — This study will use thermal forward looking infrared (FLIR) imaging to assess the severity of Complex Regional Pain Syndrome in newly diagnosed patients.

SUMMARY:
The goal of this interventional study is to explore the use of InfraRed (FLIR) imaging in determining pain intensity and severity in newly diagnosed complex regional pain syndrome patients. The main questions it aims to answer are:

Question 1: Can Infrared (FLIR) imaging be used to determine the severity of CRPS in newly diagnosed patients? Question 2: Is there any correlation with the quantification of 'the Δ thermal index value' measured by FLIR imaging with pain intensity (NRS) in newly diagnosed patients? Question 3: Is there any correlation between the quantification of 'the Δheat index value' measured by FLIR imaging between the two extremities with the severity (the severity score for CRPS) in newly diagnosed patients? Participants will have a picture of their foot taken using the forward looking infrared (FLIR) camera and answer questionnaires regarding their pain and complex regional pain syndrome (CRPS).

DETAILED DESCRIPTION:
Patients with CRPS have a better chance of remission if they receive treatment early in the disease's progression. Similarly, determining the severity of the disease early on is critical for planning effective treatment to prevent progression. The lack of an objective method for determining the severity and potential progression of CRPS is a major reason for postponing CRPS treatment.

The purpose of this interventional study is to investigate whether or not near-infrared (FLIR) imaging can be used to evaluate the level of pain experienced by patients who have recently been diagnosed with complex regional pain syndrome. Its primary goals are to provide responses to the following questions:

Question 1: Can Infrared (FLIR) imaging be used to determine the severity of CRPS in newly diagnosed patients? Question 2: Is there any correlation with the quantification of 'the Δ thermal index value' measured by FLIR imaging with pain intensity (NRS) in newly diagnosed patients? Question 3: Is there any correlation between the quantification of 'the Δheat index value' measured by FLIR imaging between the two extremities with the severity (the severity score for CRPS) in newly diagnosed patients? The forward looking infrared (FLIR) camera will be used to take a picture of each participant's foot, and they will also be asked to fill out questionnaires regarding their level of pain and complex regional pain syndrome (CRPS).

If infrared (FLIR) imaging can be used to determine the severity of CRPS in newly diagnosed patients, and if there is a correlation between the quantification of the heat index value' measured by FLIR imaging and the severity score for CRPS in newly diagnosed patients, the findings of this study could be useful in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 85 years old
* Providing CRPS diagnostic criteria using the Budapest Clinical Diagnostic Criteria.
* The patients affected with CRPS in a unilateral limb
* The patient has had pain and other symptoms for more than 3 months

Exclusion Criteria:

* Patients with suspected disc herniation, spinal stenosis, myelopathy, and suspected radiculopathy in detailed examinations and examinations (MRI, CT).
* Systemic or local infection
* Malignancy
* Pregnancy
* Uncontrollable medical and psychiatric condition
* The patients diagnosed with dysautonomia, sympathetic dysfunction(such as Raynaud disease or Buerger disease), and patients on vasoactive drugs, the mechanism of action is directly on the vasculartone.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated at the Hospital for Special Surgery for CRPS in a unilateral limb.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Complex regional pain syndrome Severity Score (CSS) | At pre-surgical screening
  The CRPS Severity Score (CSS) is a validated continuous score to measure CRPS severity. It conforms to the Budapest CRPS criteria and tracks symptoms over time. It includes 17 signs and symptoms (8 reported by the patient and 9 observed on the day of the examination). The CSS score (range 0-17) is calculated by adding reported and observed symptoms, with a higher score (17) indicating a greater number of symptoms.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) | At pre-surgical screening
  The numeric rating scale (NRS) is a pain screening tool that uses a 0-10 scale to assess pain severity at that time, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with researchers.

REFERENCES:
- [Result] Baron R, Schattschneider J, Binder A, Siebrecht D, Wasner G. Relation between sympathetic vasoconstrictor activity and pain and hyperalgesia in complex regional pain syndromes: a case-control study. Lancet. 2002 May 11;359(9318):1655-60. doi: 10.1016/S0140-6736(02)08589-6. PMID 12020526
- [Result] Bruehl S, Lubenow TR, Nath H, Ivankovich O. Validation of thermography in the diagnosis of reflex sympathetic dystrophy. Clin J Pain. 1996 Dec;12(4):316-25. doi: 10.1097/00002508-199612000-00011. PMID 8969877
- [Result] Jeon SG, Choi EJ, Lee PB, Lee YJ, Kim MS, Seo JH, Nahm FS. Do severity score and skin temperature asymmetry correlate with the subjective pain score in the patients with complex regional pain syndrome? Korean J Pain. 2014 Oct;27(4):339-44. doi: 10.3344/kjp.2014.27.4.339. Epub 2014 Oct 1. PMID 25317283
- [Result] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Schlereth T, Chont M, Vatine JJ. Development of a severity score for CRPS. Pain. 2010 Dec;151(3):870-876. doi: 10.1016/j.pain.2010.09.031. Epub 2010 Oct 20. PMID 20965657
- [Result] Krumova EK, Frettloh J, Klauenberg S, Richter H, Wasner G, Maier C. Long-term skin temperature measurements - a practical diagnostic tool in complex regional pain syndrome. Pain. 2008 Nov 15;140(1):8-22. doi: 10.1016/j.pain.2008.07.003. Epub 2008 Aug 23. PMID 18723287
- [Result] Wasner G, Schattschneider J, Baron R. Skin temperature side differences--a diagnostic tool for CRPS? Pain. 2002 Jul;98(1-2):19-26. doi: 10.1016/s0304-3959(01)00470-5. PMID 12098613

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT05852210/Prot_SAP_000.pdf